CLINICAL TRIAL: NCT06156982
Title: An Observational Study to Describe EVUSHELD™ (Tixagevimab/Cilgavimab) Pre-exposure Prophylaxis in Real-world Setting in Japan
Acronym: Evusheld DBR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8850R00032
Record Dates: First submitted 2023-11-06; First posted 2023-12-05 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; PrEP
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Evusheld administered group
  Interventions: Drug: Evusheld

INTERVENTIONS:
Drug: Evusheld — Administration of Evusheld 600 mg

SUMMARY:
This is an observational, cohort study that will use secondary data to describe the baseline demographics and clinical characteristics in patients who received EVUSHELD as PrEP against SARS-CoV-2 infection/COVID-19 in Japan.

All patients who have a record of administration of EVUSHELD in the database will be included in the study. The index date will be defined as the date of first EVUSHELD administration in the database (Day 0) and the patients will be followed up to 6 months after the index date (Day 1 to 180). The look back period is defined as the 12-month period prior to index date (Day -360 to -1). The exposure of interest will be defined as the administration of EVUSHELD for use as PrEP against COVID-19. As the result of feasibility assessment, sample size of the study expected to be approximately 280.

DETAILED DESCRIPTION:
This is an observational, cohort study that will use secondary data to describe the baseline demographics and clinical characteristics in patients who received EVUSHELD as PrEP against SARS-CoV-2 infection/COVID-19 in Japan.

All patients who have a record of administration of EVUSHELD in the database will be included in the study. The index date will be defined as the date of first EVUSHELD administration in the database (Day 0) and the patients will be followed up to 6 months after the index date (Day 1 to 180). The look back period is defined as the 12-month period prior to index date (Day -360 to -1). The exposure of interest will be defined as the administration of EVUSHELD for use as PrEP against COVID-19. As the result of feasibility assessment, sample size of the study expected to be approximately 280.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised patients who were administrated EVUSHELD as PrEP and have administration date of EVUSHELD
* patients aged ≥ 12 years at the index date

Exclusion Criteria:

* Patients who have no medical visit records at any time in the 12 months preceding the index date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have a record of administration of EVUSHELD in the database and meet the inclusion criteria and do not meet the exclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Demographics and clinical characteristics of patients received Evusheld as PrEP | Up to 360 days before the date of first administration of Evusheld
  Proportion of patients by age, gender, and clinical characteristics of interest (i.e. comorbidity, concurrent medication) between 360 days from the date of first administration of Evusheld (index date) to the index date will be described.

SECONDARY OUTCOMES:
Medically attended COVID-19 | Up to 180 days after the date of first administration of Evusheld
  Event rate and time to event for medically attended COVID-19 up to 180 days after the date of first administration of Evusheld will be described
COVID-19 hospitalization | Up to 180 days after the date of first administration of Evusheld
  Event rate and time to event for COVID-19 hospitalization up to 180 days after the date of first administration of Evusheld will be described
In-hospital mortality due to COVID-19 | Up to 180 days after the date of first administration of Evusheld
  Event rate and time to event for in-hospital mortality due to COVID-19 up to 180 days after the date of first administration of Evusheld will be described
All cause mortality | Up to 180 days after the date of first administration of Evusheld
  Event rate and time to event for all cause mortality up to 180 days after the date of first administration of Evusheld will be described

OTHER OUTCOMES:
Medically attended COVID-19 in subgroups | Up to 180 days after the date of first administration of Evusheld
  Event rate of medically attended COVID-19 by each sub groups (e.g. age, comorbidity) up to 180 days after the date of first administration of Evusheld will be described.
COVID-19 hospitalization in subgroups | Up to 180 days after the date of first administration of Evusheld
  Event rate of COVID-19 hospitalization by each sub groups (e.g. age, comorbidity) up to 180 days after the date of first administration of Evusheld will be described.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Osaka, Japan

REFERENCES:
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850R00032&attachmentIdentifier=00128184-f255-4339-9f5d-83ab1a5ad54f&fileName=D8850R00032_Evusheld_DBR_Study_report_synopsis_ver1.0.pdf&versionIdentifier=